CLINICAL TRIAL: NCT01068288
Title: Perforated Appendicitis With Delayed Presentation: Laparoscopic Appendectomy vs Expectant Management. A Randomized Clinical Trial (The PADLE Trial)
Brief Title: Perforated Appendicitis With Delayed Presentation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit adequate number of patients
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jacob Langer, Staff Surgeon, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000013658
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Appendicitis
Keywords: laparoscopic appendectomy; open appendectomy; expectant management; paediatric
MeSH Terms: conditions — Appendicitis | interventions — Laparoscopy; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Expectant Management (Experimental): Expectant Management
  Interventions: Procedure: Expectant Management
- Operative management (Experimental): Operative management
  Interventions: Procedure: Laparoscopic or open appendectomy

INTERVENTIONS:
Procedure: Laparoscopic or open appendectomy
  Arms: Operative management
Procedure: Expectant Management — A consult to Interventional Radiology will be made at the time of admission to determine whether percutaneous drainage is feasible, and if it is the abscess will be drained by Interventional Radiology. Ultrasound and/or CT scan will be used to follow the abscess collections and/or phlegmons and guide the removal of drains.
  For patients with a fecalith on imaging, a laparoscopic interval appendectomy will be performed 6-12 weeks following discharge from hospital. For those without a fecalith on imaging, a decision will be made by the family, with the guidance of the surgeon, whether or not to undergo a laparoscopic interval appendectomy.
  Arms: Expectant Management

SUMMARY:
There is no consensus among pediatric surgeons regarding the optimal treatment for children with complicated appendicitis with delayed diagnosis. With the development of broad-spectrum antibiotics, some surgeons have advocated expectant management for these children. However, there is little evidence to determine which children are most likely to benefit from this approach. Prior attempts to determine the effectiveness of expectant management for perforated appendicitis with delayed diagnosis often have not controlled for inherent differences in the clinical status of patients treated non-operatively vs. those treated with immediate appendectomy.

DETAILED DESCRIPTION:
The ability of clinical practice guidelines to improve clinical practice and optimize resource utilization continues to be substantiated in the literature. To be effective, clinical practice guidelines must be developed from reliable and reproducible data.

This trial prospectively compares expectant management versus immediate laparoscopic or open appendectomy for perforated appendicitis in children with a delayed diagnosis. The primary outcome measure is length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* All children with a delayed diagnosis of perforated appendicitis. Delayed diagnosis will be defined as symptoms for 4 or more days. Duration of symptoms will be defined as the time pain started.
* Confirmed diagnosis of perforated appendicitis. The diagnosis of perforated appendicitis will be based on diagnostic imaging (CT scan or ultrasound), showing an established appendiceal abscess or phlegmon.
* Consent to participate

Exclusion Criteria:

* Uncertainty about the diagnosis.
* The need for laparotomy for another reason.
* Free intraperitoneal air on imaging.
* Perforated appendicitis with diffuse abdominal fluid on imaging associated with a clinical picture of severe sepsis.
* Children with other medical condition that may affect the decision to operate e.g: children with inflammatory bowel disease.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Length of stay in hospital | 2 years

SECONDARY OUTCOMES:
Complications recurrent abscess, recurrent admissions related to the disease,small bowel obstruction, injury to bowel, blood loss and transfusion requirement, failure of the conservative approach | Daily until hospital discharge
Time to full parenteral intake. | Daily until hospital discharge, 6 weeks, 12 months
Duration of narcotics | Daily until hospital discharge, 6 months, 12 months
Duration of antibiotics | Daily until hospital discharge, 6 weeks, 12 months
Total dose or radiation exposure | All hospital visits until 12 months following initial discharge
Time to return to usual activity | Daily until hospital discharge, 12 months
Cost | 12 months following initial discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Langer, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada